CLINICAL TRIAL: NCT03581422
Title: Frozen-Thawed Embryo Transfers: a Comparison Between Natural Cycles With Spontaneous or Induced Ovulation
Brief Title: Natural Cycles With Spontaneous Versus Induced Ovulation in FET
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: xxxx2018
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Embryo Transfer
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NC-FET: pure natural cycle frozen-thawed embryo transfer
- mNC-FET: modified natural cycle frozen-thawed embryo transfer by hCG administration
  Interventions: Drug: hCG administration before embryo transfer

INTERVENTIONS:
Drug: hCG administration before embryo transfer — Thawed embryo transfer with ovulation triggered by hCG
  Other Names: Gonasi HP 5000 UI or Ovitrelle 250mg
  Groups: mNC-FET

SUMMARY:
In recent years, frozen-thawed embryo transfer procedure (FET) has been widely used to increase the cumulative pregnancy rate per IVF-cycle: which is the best preparation protocol remains a matter of debate.

A retrospective analysis was conducted between 2012-2017. The aim was comparing clinical pregnancy rate (CPR) of pure natural cycle frozen-thawed embryo transfer (NC-FET) versus natural cycle frozen-thawed embryo transfer with hCG-triggered ovulation (mNC-FET).

DETAILED DESCRIPTION:
Compared to repeated oocyte retrieval procedure, frozen-thawed embryo transfer (FET) has been widely used to increase the cumulative pregnancy rate per IVF-cycle, with demonstrated superiority in preventing ovarian hyperstimulation syndrome and improving cost-efficiency and time to pregnancy.

It is controversial whether triggering ovulation of the dominant follicle using human chorionic gonadotrophin (hCG) may benefit or reduce embryo implantation, when compared with a natural cycle environment. Unfavourable clinical outcomes of controlled ovarian stimulation have been reported by recently published studies, compared to the spontaneous LH surge.

This study aimed to compare the effectiveness in terms of better clinical pregnancy rates (CPR) of pure natural cycle frozen-thawed embryo transfer (NC-FET) versus natural cycle frozen-thawed embryo transfer modified by HCG administration\with hCG-triggered ovulation (mNC-FET).

A retrospective analysis was conducted between 2012-2017. In patients with regular ovulatory cycles, the timing of embryo thawing and transferring was based on spontaneous LH surge (NC-FET). Patients attended for ultrasound evaluation of the dominant follicle from Day 8 to 10 of their menstrual cycle (depending on cycle length), detecting luteinizing hormone (LH) surge in urine/ taking an ovulation test for urinary LH measurement. In selected cases, a serum assays of LH, progesterone and estradioI has been further obtained. When the endometrial thickness reached 8 mm and dominant follicle 16-20 mm in diameter, hCG was administered in absence of urinary LH surge. Embryo thawing and transfer was planned 7 days after LH surge or HCG administration, whether G5 or G6 blastocyst. Exogenous progesterone supplementation started 2 days after hCG administration versus the same day of embryo transfer procedure in NC- ET. To limit potential confounders, only single blastocyst transfer cycles were included, vitrified on Days 5 or 6, excluding PGT-a (Pre Gestational Test for aneuploydia) cycles and cleavage stage embryo transfers. A unilevel and multi level logistic regression analysis was conducted using Stata Software versione15.

ELIGIBILITY:
Inclusion Criteria:

* only single blastocyst transfer cycles were included

Exclusion Criteria:

* PGT-a cycles and cleavage stage embryo transfers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 2866 cycles were included in the analysis. To limit potential confounders, only single blastocyst transfer cycles were included, vitrified on Days 5 or 6, excluding PGT-a cycles and cleavage stage embryo transfers.
Sampling Method: Non-Probability Sample
Enrollment: 2866 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
CPR in NCFET vs mNCFET | 2012-2017
  compare the effectiveness in terms of better clinical pregnancy rates (CPR) of pure natural cycle frozen-thawed embryo transfer (NC-FET) versus natural cycle frozen-thawed embryo transfer modified by HCG administration

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levi Setti PE, Cirillo F, De Cesare R, Morenghi E, Canevisio V, Ronchetti C, Baggiani A, Smeraldi A, Albani E, Patrizio P. Seven Years of Vitrified Blastocyst Transfers: Comparison of 3 Preparation Protocols at a Single ART Center. Front Endocrinol (Lausanne). 2020 May 29;11:346. doi: 10.3389/fendo.2020.00346. eCollection 2020. PMID 32547496